CLINICAL TRIAL: NCT02719171
Title: A Randomised, Double-blind, Placebo-controlled, Proof-of-concept, Dose-ranging Study of BI 655066/ABBV-066/Risankizumab in Patients With Active Psoriatic Arthritis
Brief Title: BI 655066/ABBV-066/Risankizumab Compared to Placebo in Patients With Active Psoriatic Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M16-002; 2015-003625-34 (EudraCT Number); 1311.5 (Other: Boehringer Ingelheim)
Record Dates: First submitted 2016-03-18; First posted 2016-03-25 (Estimated); Results first posted 2019-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Arthritis, Psoriatic
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — risankizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator): Participants randomized to receive double-blind (DB) placebo for risankizumab by subcutaneous (SC) injection every 4 weeks for 16 weeks.
  Interventions: Drug: placebo for risankizumab
- Risankizumab 150 mg Every 4 Weeks (Experimental): Participants randomized to receive double-blind (DB) risankizumab 150 mg by subcutaneous (SC) injection every 4 weeks for 16 weeks.
  Interventions: Drug: risankizumab
- Risankizumab 150 mg Weeks 0, 4, and 16 (Experimental): Participants randomized to receive double-blind (DB) risankizumab 150 mg by subcutaneous (SC) injection at Weeks 0, 4, and 16.
  Interventions: Drug: risankizumab
- Risankizumab 150 mg Weeks 0 and 12 (Experimental): Participants randomized to receive double-blind (DB) risankizumab 150 mg by subcutaneous (SC) injection at Weeks 0 and 12.
  Interventions: Drug: risankizumab
- Risankizumab 75 mg Week 0 (Experimental): Participants randomized to receive double-blind (DB) risankizumab 75 mg by subcutaneous (SC) injection at Week 0.
  Interventions: Drug: risankizumab

INTERVENTIONS:
Drug: risankizumab — Risankizumab administered by SC injection
  Other Names: BI 655066; ABBV-066; SKYRIZI
  Arms: Risankizumab 150 mg Every 4 Weeks; Risankizumab 150 mg Weeks 0 and 12; Risankizumab 150 mg Weeks 0, 4, and 16; Risankizumab 75 mg Week 0
Drug: placebo for risankizumab — Placebo for risankizumab administered by SC injection
  Arms: Placebo

SUMMARY:
The overall purpose of this trial is to assess clinical efficacy and safety of different subcutaneous doses of BI 655066/ABBV-066/risankizumab in adult patients with psoriatic arthritis in order to select doses for further clinical trials.

ELIGIBILITY:
Inclusion criteria:

* Have psoriatic arthritis (PsA) symptoms for ≥ 6 months prior to screening, as assessed by the investigator
* Have PsA on the basis of the Classification Criteria for Psoriatic Arthritis (CASPAR) with peripheral symptoms at screening visit, as assessed by the investigator
* Have ≥ 5 tender joints and ≥ 5 swollen joints at screening and randomisation visits, as assessed by the investigator
* At least one psoriasis (PsO) lesion or a documented personal history of PsO at screening, as assessed by the investigator
* If patients receive concurrent PsA treatments, these need to be on stable doses
* Active PsA that has been inadequately controlled by standard doses of non-steroidal anti-inflammatory drugs (NSAIDs) administered for ≥ 4 weeks, or traditional disease-modifying anti-rheumatic drugs (DMARDs) (including sulfasalazine) administered for ≥ 3 months, or tumor necrosis factor inhibitor (TNFi) agents, or subjects are intolerant to NSAIDs or DMARDs or tumor necrosis factor inhibitor (TNFi) agents, as assessed by the investigator

Exclusion criteria:

* Major chronic inflammatory or connective tissue disease other than PsA (e.g. rheumatoid arthritis, systemic lupus erythematosus, ankylosing spondylitis, Lyme disease, gout) and fibromyalgia, as assessed by the investigator
* Has received any therapeutic agent directly targeted to interleukin 12/23 (IL-12/23) (including ustekinumab), IL-23 or IL-17 (including secukinumab)
* Prior use of more than two different TNFi agents
* Use of the following treatments: TNFi agents within 12 weeks, etanercept within 8 weeks, leflunomide without cholestyramine wash-out within 8 weeks, systemic non-biologic medications for psoriatic arthritis or psoriasis and photochemotherapy within 4 weeks, intraarticular injections (including steroids) and intramuscular or intravenous corticosteroid treatment within 4 weeks, topical psoriasis medications and phototherapy within 2 weeks, low and high potency opioid analgesics within 2 weeks prior to randomisation
* Plans for administration of live vaccines during the study period or within 6 weeks prior to randomisation
* History of allergy/hypersensitivity to a systemically administered biologic agent or its excipients
* Active systemic infections during the last 2 weeks (exception: common cold) prior to randomisation, as assessed by the investigator
* Chronic or relevant acute infections including HIV, viral hepatitis and (or) active tuberculosis (TB). Patients with a positive QuantiFERON TB or purified protein derivate (PPD) test may participate in the study if further work up (according to local practice/guidelines) establishes conclusively that the patient has no evidence of active TB.
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal or squamous cell carcinoma of the skin or in situ carcinoma of uterine cervix
* Major surgery performed within 12 weeks prior to randomisation or planned within 32 weeks after randomisation (e.g. hip replacement, aneurysm removal, stomach ligation), as assessed by the investigator
* Total white blood count (WBC) < 3,000/µL, or platelets < 100,000/µL or neutrophils < 1,500/µL, or hemoglobin < 8.5 g/dL at screening
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2x the upper limit of normal, or serum direct bilirubin ≥ 1.5 mg/dL at screening
* Positive rheumatoid factor or anti-cyclic-citrullinated peptide (anti-CCP) antibodies at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim

REFERENCES:
- [Derived] Thakre N, D'Cunha R, Goebel A, Liu W, Pang Y, Suleiman AA. Population Pharmacokinetics and Exposure-Response Analyses for Risankizumab in Patients with Active Psoriatic Arthritis. Rheumatol Ther. 2022 Dec;9(6):1587-1603. doi: 10.1007/s40744-022-00495-0. Epub 2022 Sep 30. PMID 36178584
- [Derived] Mease PJ, Kellner H, Morita A, Kivitz AJ, Aslanyan S, Padula SJ, Topp AS, Eldred A, Behrens F, Papp KA. Long-Term Efficacy and Safety of Risankizumab in Patients with Active Psoriatic Arthritis: Results from a 76-Week Phase 2 Randomized Trial. Rheumatol Ther. 2022 Oct;9(5):1361-1375. doi: 10.1007/s40744-022-00474-5. Epub 2022 Aug 5. PMID 35931879
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included a 6-week screening period.
Period: Overall Study
Arm/Group | Placebo | Risankizumab 150 mg Every 4 Weeks | Risankizumab 150 mg Weeks 0, 4, and 16 | Risankizumab 150 mg Weeks 0 and 12 | Risankizumab 75 mg Week 0
Started | 42 | 42 | 42 | 39 | 20
Completed | 41 | 38 | 39 | 37 | 18
Not Completed | 1 | 4 | 3 | 2 | 2
Not completed — Adverse Event | 1 | 2 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0
Not completed — Subject Withdrawal | 0 | 2 | 2 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All randomized participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Risankizumab 150 mg Every 4 Weeks | Risankizumab 150 mg Weeks 0, 4, and 16 | Risankizumab 150 mg Weeks 0 and 12 | Risankizumab 75 mg Week 0 | Total
Number analyzed (Participants) | 42 | 42 | 42 | 39 | 20 | 185
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (11.16) | 51.8 (14.56) | 50.1 (12.33) | 51.6 (11.87) | 53.8 (10.98) | 51.0 (12.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 14 | 17 | 10 | 80
  Male | 24 | 21 | 28 | 22 | 10 | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 0 | 0 | 3
  Not Hispanic or Latino | 40 | 41 | 39 | 38 | 19 | 177
  Unknown or Not Reported | 0 | 1 | 2 | 1 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 5 | 6 | 3 | 4 | 4 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 36 | 35 | 37 | 34 | 15 | 157
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 2 | 1 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response at Week 16
Description: Response defined by ACR20 criteria (improvement from baseline) at Week 16: ≥ 20% improvement in tender joint count; ≥ 20% improvement in swollen joint count; and ≥ 20% improvement in at least 3 of the 5 following parameters:
  * Patient assessment of pain
  * Patient global assessment of disease activity
  * Investigator's global assessment of disease activity
  * Health Assessment Questionnaire Disability Index (HAQ-DI)
  * Acute phase reactant value (C-reactive protein).
  Nonresponder imputation (NRI) was used for missing data.
Time Frame: Week 16
Population: FAS
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Risankizumab 150 mg Every 4 Weeks; 150 mg Weeks 0, 4, 16: Participants randomized to receive double-blind (DB) risankizumab 150 mg by subcutaneous (SC) injection every 4 weeks for 16 weeks AND participants randomized to receive DB risankizumab 150 mg by SC injection at Weeks 0, 4, and 16.
- Risankizumab 150 mg Weeks 0, 4, and 16; 150 mg Weeks 0 and 12: Participants randomized to receive double-blind (DB) risankizumab 150 mg by subcutaneous (SC) injection at Weeks 0, 4, and 16 AND participants randomized to receive double-blind (DB) risankizumab 150 mg by subcutaneous (SC) injection at Weeks 0 and 12.
Arm/Group | Placebo | Risankizumab 150 mg Every 4 Weeks | Risankizumab 150 mg Weeks 0, 4, and 16 | Risankizumab 150 mg Weeks 0 and 12 | Risankizumab 75 mg Week 0 | Risankizumab 150 mg Every 4 Weeks; 150 mg Weeks 0, 4, 16 | Risankizumab 150 mg Weeks 0, 4, and 16; 150 mg Weeks 0 and 12
Number analyzed (Participants) | 42 | 42 | 42 | 39 | 20 | 84 | 81
percentage of participants | 35.7 [23.5 to 49.5] | 57.1 [43.3 to 70.2] | 61.9 [48.0 to 74.4] | 59.0 [44.6 to 72.3] | 65.0 [44.2 to 82.3] | 59.5 [50.0 to 68.6] | 60.5 [50.8 to 69.6]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 150 mg Every 4 Weeks; 150 mg Weeks 0, 4, 16; The 90% confidence interval (CI) for the difference in response rates between the groups and the 2-sided p-value are calculated using the Cochran Mantel-Haenszel method, stratified by prior tumor necrosis factor inhibitor (TNFi) use and concurrent methotrexate use; Test type: Other; p = 0.007, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 24.0, 90% CI 2-sided [9.3 to 38.7]

2. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Response at Week 16
Description: Response defined by ACR50 criteria (improvement from baseline) at Week 16: ≥ 50% improvement in tender joint count; ≥ 50% improvement in swollen joint count; and ≥ 50% improvement in at least 3 of the 5 following parameters:
  * Patient assessment of pain
  * Patient global assessment of disease activity
  * Investigator's global assessment of disease activity
  * HAQ-DI
  * Acute phase reactant value (C-reactive protein).
  NRI was used for missing data.
Time Frame: Week 16
Population: FAS
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Risankizumab 150 mg Every 4 Weeks; 150 mg Weeks 0, 4, and 16: Participants randomized to receive double-blind (DB) risankizumab 150 mg by subcutaneous (SC) injection every 4 weeks for 16 weeks AND participants randomized to receive DB risankizumab 150 mg by SC injection at Weeks 0, 4, and 16.
Arm/Group | Placebo | Risankizumab 150 mg Every 4 Weeks | Risankizumab 150 mg Weeks 0, 4, and 16 | Risankizumab 150 mg Weeks 0 and 12 | Risankizumab 75 mg Week 0 | Risankizumab 150 mg Every 4 Weeks; 150 mg Weeks 0, 4, and 16 | Risankizumab 150 mg Weeks 0, 4, and 16; 150 mg Weeks 0 and 12
Number analyzed (Participants) | 42 | 42 | 42 | 39 | 20 | 84 | 81
percentage of participants | 11.9 [4.8 to 23.4] | 23.8 [13.5 to 37.0] | 23.8 [13.5 to 37.0] | 38.5 [25.4 to 52.9] | 25.0 [10.4 to 45.6] | 23.8 [16.4 to 32.7] | 30.9 [22.5 to 40.4]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 150 mg Every 4 Weeks; 150 mg Weeks 0, 4, and 16; The 90% CI for the difference in response rates between the groups and the 2-sided p-value are calculated using the Cochran Mantel-Haenszel method, stratified by prior TNFi use and concurrent methotrexate use; Test type: Other; p = 0.074, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 12.0, 90% CI 2-sided [1.0 to 23.0]
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 150 mg Weeks 0, 4, and 16; 150 mg Weeks 0 and 12; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.007, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 19.0, 90% CI 2-sided [7.4 to 30.6]

3. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Response at Week 16
Description: Response defined by ACR70 criteria (improvement from baseline) at Week 16: ≥ 70% improvement in tender joint count; ≥ 70% improvement in swollen joint count; and ≥ 70% improvement in at least 3 of the 5 following parameters:
  * Patient assessment of pain
  * Patient global assessment of disease activity
  * Investigator's global assessment of disease activity
  * HAQ-DI
  * Acute phase reactant value (C-reactive protein).
  NRI was used for missing data.
Time Frame: Week 16
Population: FAS
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab 150 mg Every 4 Weeks | Risankizumab 150 mg Weeks 0, 4, and 16 | Risankizumab 150 mg Weeks 0 and 12 | Risankizumab 75 mg Week 0 | Risankizumab 150 mg Every 4 Weeks; 150 mg Weeks 0, 4, and 16 | Risankizumab 150 mg Weeks 0, 4, and 16; 150 mg Weeks 0 and 12
Number analyzed (Participants) | 42 | 42 | 42 | 39 | 20 | 84 | 81
percentage of participants | 0.0 [0.0 to 6.9] | 14.3 [6.4 to 26.3] | 7.1 [2.0 to 17.4] | 25.6 [14.6 to 39.6] | 15.0 [4.2 to 34.4] | 10.7 [5.7 to 18.0] | 16.0 [9.8 to 24.3]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 150 mg Every 4 Weeks; 150 mg Weeks 0, 4, and 16; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.006, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 10.3, 90% CI 2-sided [4.1 to 16.4]
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 150 mg Weeks 0, 4, and 16; 150 mg Weeks 0 and 12; [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 15.7, 90% CI 2-sided [8.5 to 22.9]

4. Secondary Outcome: Tender Joint Count (TJC68): Change From Baseline to Week 16
Description: Sixty-eight joints were assessed and classified as either tender (1) or not tender (0). A negative change represents a decrease in the number of tender joints.
Time Frame: Baseline, Week 16
Population: Participants in the FAS with available data at Baseline and Week 16.
Measure: Least Squares Mean (90% Confidence Interval); unit: tender joints
Arm/Group | Placebo | Risankizumab 150 mg Every 4 Weeks | Risankizumab 150 mg Weeks 0, 4, and 16 | Risankizumab 150 mg Weeks 0 and 12 | Risankizumab 75 mg Week 0 | Risankizumab 150 mg Every 4 Weeks; 150 mg Weeks 0, 4, and 16 | Risankizumab 150 mg Weeks 0, 4, and 16; 150 mg Weeks 0 and 12
Number analyzed (Participants) | 42 | 40 | 41 | 38 | 18 | 81 | 79
tender joints | -7.9 [-10.6 to -5.2] | -7.8 [-10.6 to -5.1] | -9.6 [-12.4 to -6.9] | -10.4 [-13.2 to -7.5] | -10.8 [-14.9 to -6.8] | -8.6 [-10.5 to -6.6] | -9.9 [-11.8 to -8.0]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 150 mg Every 4 Weeks; 150 mg Weeks 0, 4, and 16; The 2-sided p-value is calculated using a mixed model repeated measures model with categorical fixed effects of treatment, stratification factors, week, and treatment-by-week interaction and the continuous fixed baseline measurement, with subject as a random effect; Test type: Other; p = 0.690, mixed model repeated measures model; Mean Difference (Final Values) = -0.8, 90% CI 2-sided [-4.0 to 2.5]
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 150 mg Weeks 0, 4, and 16; 150 mg Weeks 0 and 12; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.260, mixed model repeated measures model; Mean Difference (Final Values) = -2.1, 90% CI 2-sided [-5.3 to 1.0]

5. Secondary Outcome: Swollen Joint Count (SJC): Change From Baseline to Week 16
Description: Sixty-six joints were assessed and classified as either swollen (1) or not swollen (0). A negative change represents a decrease in the number of tender joints.
Time Frame: Baseline, Week 16
Population: Participants in the FAS with available data at Baseline and Week 16.
Measure: Least Squares Mean (90% Confidence Interval); unit: swollen joints
Arm/Group | Placebo | Risankizumab 150 mg Every 4 Weeks | Risankizumab 150 mg Weeks 0, 4, and 16 | Risankizumab 150 mg Weeks 0 and 12 | Risankizumab 75 mg Week 0 | Risankizumab 150 mg Every 4 Weeks; 150 mg Weeks 0, 4, and 16 | Risankizumab 150 mg Weeks 0, 4, and 16; 150 mg Weeks 0 and 12
Number analyzed (Participants) | 42 | 40 | 41 | 38 | 18 | 81 | 79
swollen joints | -7.1 [-8.5 to -5.7] | -6.8 [-8.3 to -5.4] | -7.8 [-9.3 to -6.4] | -8.3 [-9.7 to -6.8] | -7.8 [-9.9 to -5.7] | -7.3 [-8.5 to -6.2] | -8.3 [-9.4 to -7.2]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 150 mg Every 4 Weeks; 150 mg Weeks 0, 4, and 16; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.791, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -0.3, 90% CI 2-sided [-2.1 to 1.5]
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 150 mg Weeks 0, 4, and 16; 150 mg Weeks 0 and 12; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.320, mixed model repeated measures model; Mean Difference (Final Values) = -1.1, 90% CI 2-sided [-2.8 to 0.7]

6. Secondary Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI) Score: Change From Baseline to Week 16
Description: The HAQ-DI is a patient-reported questionnaire specific for rheumatoid arthritis that consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 very severe, high-dependency disability. HAQ remission indicating normal physical function is defined by HAQ-DI score of < 0.5. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Week 16
Population: Participants in the FAS with available data at Baseline and Week 16.
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Risankizumab 150 mg Every 4 Weeks | Risankizumab 150 mg Weeks 0, 4, and 16 | Risankizumab 150 mg Weeks 0 and 12 | Risankizumab 75 mg Week 0 | Risankizumab 150 mg Every 4 Weeks; 150 mg Weeks 0, 4, and 16 | Risankizumab 150 mg Weeks 0, 4, and 16; 150 mg Weeks 0 and 12
Number analyzed (Participants) | 42 | 39 | 40 | 38 | 18 | 79 | 78
units on a scale | -0.089 [-0.204 to 0.026] | -0.182 [-0.299 to -0.065] | -0.163 [-0.280 to -0.047] | -0.245 [-0.365 to -0.126] | -0.147 [-0.317 to 0.023] | -0.184 [-0.270 to -0.099] | -0.206 [-0.291 to -0.120]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 150 mg Every 4 Weeks; 150 mg Weeks 0, 4, and 16; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.341, mixed model repeated measures model; mixed model repeated measures model = -0.082, 90% CI 2-sided [-0.225 to 0.060]
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 150 mg Weeks 0, 4, and 16; 150 mg Weeks 0 and 12; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.181, mixed model repeated measures model; Mean Difference (Final Values) = -0.114, 90% CI 2-sided [-0.254 to 0.027]

7. Secondary Outcome: Short Form-36 Health Status Survey (SF-36) Physical Component: Change From Baseline to Week 16
Description: The SF-36 determined participant's overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 comprise the physical component of the SF-36. Scores on each item were summed and averaged (range = 0-100); a positive change from Baseline indicates improvement.
Time Frame: Baseline, Week 16
Population: Participants in the FAS with available data at Baseline and Week 16.
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Risankizumab 150 mg Every 4 Weeks | Risankizumab 150 mg Weeks 0, 4, and 16 | Risankizumab 150 mg Weeks 0 and 12 | Risankizumab 75 mg Week 0 | Risankizumab 150 mg Every 4 Weeks; 150 mg Weeks 0, 4, and 16 | Risankizumab 150 mg Weeks 0, 4, and 16; 150 mg Weeks 0 and 12
Number analyzed (Participants) | 42 | 37 | 41 | 39 | 19 | 78 | 80
units on a scale | 1.93 [0.17 to 3.70] | 3.87 [2.03 to 5.71] | 3.50 [1.72 to 5.27] | 3.10 [1.27 to 4.93] | 7.42 [4.81 to 10.03] | 3.80 [2.52 to 5.08] | 3.32 [2.03 to 4.62]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 150 mg Every 4 Weeks; 150 mg Weeks 0, 4, and 16; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.174, mixed model repeated measures model; Mean Difference (Final Values) = 1.70, 90% CI 2-sided [-0.36 to 3.77]
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 150 mg Weeks 0, 4, and 16; 150 mg Weeks 0 and 12; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.284, mixed model repeated measures model; Mean Difference (Final Values) = 1.35, 90% CI 2-sided [-0.73 to 3.44]

8. Secondary Outcome: SF-36 Mental Component: Change From Baseline to Week 16
Description: The SF-36 determined participant's overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 5-8 comprise the mental component of the SF-36. Scores on each item were summed and averaged (range = 0-100); a positive change from Baseline indicates improvement.
Time Frame: Baseline, Week 16
Population: Participants in the FAS with available data at Baseline and Week 16.
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Risankizumab 150 mg Every 4 Weeks | Risankizumab 150 mg Weeks 0, 4, and 16 | Risankizumab 150 mg Weeks 0 and 12 | Risankizumab 75 mg Week 0 | Risankizumab 150 mg Every 4 Weeks; 150 mg Weeks 0, 4, and 16 | Risankizumab 150 mg Weeks 0, 4, and 16; 150 mg Weeks 0 and 12
Number analyzed (Participants) | 42 | 37 | 41 | 39 | 19 | 78 | 80
units on a scale | 0.48 [-1.74 to 2.69] | -0.36 [-2.68 to 1.96] | 2.26 [0.03 to 4.49] | 2.84 [0.54 to 5.14] | -1.08 [-4.35 to 2.19] | 1.31 [-0.38 to 3.00] | 2.29 [0.59 to 3.99]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 150 mg Every 4 Weeks; 150 mg Weeks 0, 4, and 16; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.718, mixed model repeated measures model; Mean Difference (Final Values) = 0.59, 90% CI 2-sided [-2.12 to 3.30]
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 150 mg Weeks 0, 4, and 16; 150 mg Weeks 0 and 12; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.204, mixed model repeated measures model; Mean Difference (Final Values) = 2.06, 90% CI 2-sided [-0.61 to 4.74]

9. Secondary Outcome: Dactylitis Count: Change From Baseline to Week 16 in Participants With Dactylitis at Baseline
Description: The number of fingers and toes with dactylitis (ranging from 0 to 20). A negative change represents a decrease in the number of fingers and toes affected by dactylitis.
Time Frame: Baseline, Week 16
Population: Participants in the FAS with available data at Baseline and Week 16.
Measure: Least Squares Mean (90% Confidence Interval); unit: fingers and toes with dactylitis
Arm/Group | Placebo | Risankizumab 150 mg Every 4 Weeks | Risankizumab 150 mg Weeks 0, 4, and 16 | Risankizumab 150 mg Weeks 0 and 12 | Risankizumab 75 mg Week 0 | Risankizumab 150 mg Every 4 Weeks; 150 mg Weeks 0, 4, and 16 | Risankizumab 150 mg Weeks 0, 4, and 16; 150 mg Weeks 0 and 12
Number analyzed (Participants) | 9 | 11 | 11 | 10 | 5 | 22 | 21
fingers and toes with dactylitis | -2.6 [-3.9 to -1.4] | -1.1 [-2.2 to 0.1] | -1.9 [-3.0 to -0.8] | -2.9 [-4.1 to -1.7] | -3.5 [-5.2 to -1.8] | -1.5 [-2.4 to -0.6] | -2.4 [-3.0 to -1.9]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 150 mg Every 4 Weeks; 150 mg Weeks 0, 4, and 16; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.243, mixed model repeated measures model; Mean Difference (Final Values) = 1.2, 90% CI 2-sided [-0.5 to 2.8]
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 150 mg Weeks 0, 4, and 16; 150 mg Weeks 0 and 12; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.906, mixed model repeated measures model; Mean Difference (Final Values) = 0.1, 90% CI 2-sided [-1.0 to 1.1]

10. Secondary Outcome: Spondyloarthritis Research Consortium of Canada (SPARCC) Enthesitis Index: Change From Baseline to Week 16 in Participants With Enthesitis at Baseline
Description: Assessment of enthesitis was performed in the following 16 domains: left and right (L/R) medial epicondyle; L/R lateral epicondyle; L/R supraspinatus insertion into the greater tuberosity of humerus; L/R greater trochanter; L/R quadriceps insertion into superior border of patella; L/R patellar ligament insertion into inferior pole of patella or tibial tubercle; L/R Achilles tendon insertion into calcaneum; L/R plantar fascia insertion into calcaneum. Tenderness at each site was classified as either absent (0) or present (1) to yield total SPARCC scores ranging from 0 (0 sites with tenderness) to 16 (16 sites with tenderness). A negative change from Baseline indicates improvement.
Time Frame: Baseline, Week 16
Population: Participants in the FAS with enthesitis at Baseline and with available data at Baseline and Week 16.
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Risankizumab 150 mg Every 4 Weeks | Risankizumab 150 mg Weeks 0, 4, and 16 | Risankizumab 150 mg Weeks 0 and 12 | Risankizumab 75 mg Week 0 | Risankizumab 150 mg Every 4 Weeks; 150 mg Weeks 0, 4, and 16 | Risankizumab 150 mg Weeks 0, 4, and 16; 150 mg Weeks 0 and 12
Number analyzed (Participants) | 27 | 27 | 24 | 25 | 11 | 51 | 49
units on a scale | -1.1 [-2.1 to -0.2] | -1.4 [-2.3 to -0.5] | -2.4 [-3.3 to -1.4] | -1.8 [-2.7 to -0.8] | -3.7 [-5.1 to -2.3] | -1.7 [-2.4 to -1.0] | -2.1 [-2.7 to -1.4]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 150 mg Every 4 Weeks; 150 mg Weeks 0, 4, and 16; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.325, mixed model repeated measures model; Mean Difference (Final Values) = -0.7, 90% CI 2-sided [-1.8 to 0.5]
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 150 mg Weeks 0, 4, and 16; 150 mg Weeks 0 and 12; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.160, mixed model repeated measures model; Mean Difference (Final Values) = -0.9, 90% CI 2-sided [-2.1 to 0.2]

11. Secondary Outcome: Modified Nail Psoriasis Severity Index (mNAPSI): Change From Baseline to Week 16
Description: mNAPSI grades each fingernail for onycholysis (separation of the nail plate from the nail bed) and oil-drop (salmon patch) dyschromia (reddish-brown discoloration under the nail plate) on a scale of 0 (none present) to 3 (>30% of the nail); pitting (small, sharply defined depressions in the nail surface) on a scale of 0 (0 pits present) to 3 (>50 pits present); nail plate crumbling on a scale of 0 (no crumbling) to 3 (>50% of nail has crumbling); and presence (1) or absence (0) of leukonychia (white spots), splinter hemorrhages, nail bed hyperkeratosis, and red spots in the lunula. mNAPSI is calculated as the sum of all the components for all of the participants fingernails, for a minimal - maximal total score of 0 to 130. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Week 16
Population: Participants in the FAS with enthesitis at Baseline and with available data at Baseline and Week 16.
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Risankizumab 150 mg Every 4 Weeks | Risankizumab 150 mg Weeks 0, 4, and 16 | Risankizumab 150 mg Weeks 0 and 12 | Risankizumab 75 mg Week 0 | Risankizumab 150 mg Every 4 Weeks; 150 mg Weeks 0, 4, and 16 | Risankizumab 150 mg Weeks 0, 4, and 16; 150 mg Weeks 0 and 12
Number analyzed (Participants) | 28 | 19 | 23 | 25 | 9 | 42 | 48
units on a scale | -5.2 [-7.4 to -3.0] | -6.7 [-9.4 to -4.1] | -5.8 [-8.2 to -3.4] | -10.7 [-13.1 to -8.3] | -6.8 [-10.6 to -3.0] | -5.5 [-7.3 to -3.8] | -8.1 [-9.9 to -6.3]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 150 mg Every 4 Weeks; 150 mg Weeks 0, 4, and 16; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.453, mixed model repeated measures model; Mean Difference (Final Values) = -1.2, 90% CI 2-sided [-4.0 to 1.5]
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 150 mg Weeks 0, 4, and 16; 150 mg Weeks 0 and 12; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.111, mixed model repeated measures model; Mean Difference (Final Values) = -2.8, 90% CI 2-sided [-5.7 to 0.1]

12. Secondary Outcome: Percentage of Participants Achieving 90% Improvement in Psoriasis Area and Severity Index (PASI) Score (PASI90) at Week 16
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI90 is defined as at least a 90% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100. The percentage of participants achieving PASI90 at Week 16 are provided. NRI was used for missing data.
Time Frame: Week 16
Population: FAS
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab 150 mg Every 4 Weeks | Risankizumab 150 mg Weeks 0, 4, and 16 | Risankizumab 150 mg Weeks 0 and 12 | Risankizumab 75 mg Week 0 | Risankizumab 150 mg Every 4 Weeks; 150 mg Weeks 0, 4, and 16 | Risankizumab 150 mg Weeks 0, 4, and 16; 150 mg Weeks 0 and 12
Number analyzed (Participants) | 21 | 12 | 18 | 23 | 9 | 30 | 41
percentage of participants | 9.5 [1.7 to 27.1] | 58.3 [31.5 to 81.9] | 66.7 [44.6 to 84.4] | 52.2 [33.5 to 70.4] | 55.6 [25.1 to 83.1] | 63.3 [46.7 to 77.9] | 58.5 [44.5 to 71.6]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 150 mg Every 4 Weeks; 150 mg Weeks 0, 4, and 16; [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 53.5, 90% CI 2-sided [35.9 to 71.1]
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 150 mg Weeks 0, 4, and 16; 150 mg Weeks 0 and 12; [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 48.8, 90% CI 2-sided [33.1 to 64.5]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug until 15 weeks after the last dose of study drug (up to 31 weeks).
Arm/Group | Placebo | Risankizumab 150 mg Every 4 Weeks | Risankizumab 150 mg Weeks 0, 4, and 16 | Risankizumab 150 mg Weeks 0 and 12 | Risankizumab 75 mg Week 0
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42 | 0/42 | 0/39 | 0/20
Serious Adverse Events (participants affected / at risk) | 2/42 | 3/42 | 0/42 | 2/39 | 3/20
Other Adverse Events (participants affected / at risk) | 25/42 | 16/42 | 13/42 | 19/39 | 13/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=42) | Risankizumab 150 mg Every 4 Weeks (N=42) | Risankizumab 150 mg Weeks 0, 4, and 16 (N=42) | Risankizumab 150 mg Weeks 0 and 12 (N=39) | Risankizumab 75 mg Week 0 (N=20)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal septal operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=42) | Risankizumab 150 mg Every 4 Weeks (N=42) | Risankizumab 150 mg Weeks 0, 4, and 16 (N=42) | Risankizumab 150 mg Weeks 0 and 12 (N=39) | Risankizumab 75 mg Week 0 (N=20)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 2 (2) | 3 (6) | 2 (2) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 7 (12) | 5 (6) | 9 (11) | 4 (6)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 3 (3) | 3 (3) | 1 (2) | 3 (4) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2016-10-12): https://cdn.clinicaltrials.gov/large-docs/71/NCT02719171/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/71/NCT02719171/SAP_001.pdf